CLINICAL TRIAL: NCT04808947
Title: The Ideal Analgesic Technique for Total Knee Arthroplasty: A Randomized Comparison Between Local Infiltration Analgesia Alone or Combined With Adductor Canal and iPACK Blocks
Brief Title: LIA vs. LIA + ACB-iPACK Block for Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LIA vs. LIA + ACB-iPACK block
Record Dates: First submitted 2021-03-08; First posted 2021-03-22 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Nerve Block; Neuromuscular Blockade

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group, triple blind (patient, assessor, anesthesiologist in the operating room)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local infiltration analgesia (Experimental): Patients in this group will receive LIA intraoperatively, as per institutional standard. The injected solution will be comprised of 100cc Ropiv 2%, + Ketorolac 30 mg + Epinephrine 25 ug.
  Interventions: Procedure: Local infiltration analgesia
- Local infiltration analgesia + ACB-iPACK block (Active Comparator): Patients in this group will receive LIA intraoperatively, as per institutional standard. The injected solution will be comprised of 100cc Ropiv 2%, + Ketorolac 30 mg + Epinephrine 25 ug.
  Patients in this group will also receive preoperative nerve blocks under ultrasound guidance. These will include:
  1. Adductor canal block with 0.5% Ropivacaine w/epi 20 mL
  2. iPack block with 0.25% Ropivacaine w/epi 10 mL
  Interventions: Procedure: Local infiltration analgesia; Procedure: Ultrasound-guided adductor canal block

INTERVENTIONS:
Procedure: Local infiltration analgesia — Procedure: Local infiltration analgesia performed by surgeons.
Procedure: Ultrasound-guided adductor canal block — Procedure: Ultrasound-guided adductor canal and iPACK blocks performed by anesthesiologists preoperatively.
  Other Names: iPACK block
  Arms: Local infiltration analgesia + ACB-iPACK block

SUMMARY:
LIA is the mainstay of postoperative analgesia in patients having knee arthroplasty. The combination of ACB-iPACK blocks has also been proposed as an effective analgesic modality for total knee arthroplasty. However, whether combining these two modalities yields any important incremental analgesic benefit remains unclear. The investigators hypothesized that the addition of ACB and iPACK blocks to LIA will yield clinically important analgesic benefits compared to LIA alone in patients having total knee arthroplasty.

DETAILED DESCRIPTION:
LIA is the mainstay of postoperative analgesia in patients having knee arthroplasty. Performed by surgeons, LIA provides effective postoperative pain relief and reduces opioid requirements. Similar analgesic benefits have also been attributed to adductor canal and iPACK blocks, which partially block sensory innervation to the knee and its posterior capsule. Performed by anesthesiologist preoperatively, these blocks have also been incorporated into the care standard in numerous centers. However, it is not clear whether adding the adductor canal and iPACK blocks yields any incremental analgesic benefits. The investigators aimed to evaluate the benefits of adding adductor canal and iPACK blocks to LIA in patients having total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. ASA classification I-III
2. BMI < 35 kg/m2
3. Having elective unilateral total knee arthroplasty

Exclusion Criteria:

1. Bilateral knee surgery.
2. Pre-existing neurological deficit or peripheral neuropathy in the lower the lower limbs
3. Severe, poorly controlled cardiac conditions, significant arrhythmias, severe valvular heart diseases
4. Severe, poorly controlled respiratory conditions (severe COPD, severe interstitial lung disease, severe / poorly controlled asthma)
5. Contraindication to regional anesthesia (e.g. bleeding diathesis, coagulopathy, sepsis, infection at the site of potential needle puncture on the posterior chest)
6. Patient refusal
7. Chronic pain disorder
8. Chronic opioid use (≥30 mg oxycodone / day)
9. Contraindication (or allergy) to a component of multi-modal analgesia protocol
10. Allergy to amide local anesthetics used in nerve blocks
11. Contraindications to spinal anesthesia
12. Significant psychiatric disorder that would preclude objective study assessment
13. Pregnancy
14. Inability to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain at rest | over the first 24 hours
  Area under the curve
Quality of recovery (QoR-15) | 24 hours postoperatively
  Quality of Recovery (QR15) scores at 24 hours will be the second primary outcome.
  QR15 is a measurement of quality of recovery after surgery and anesthesia that has been psychometrically tested and validated. Reporting of outcome measures on a scale of 0 to 10 (0=None of the time and 10=All of the time). There are a total of 40 items/questions.

SECONDARY OUTCOMES:
Mean opioid analgesic consumption | 24 hours postoperatively
  Postoperative cumulative oral morphine equivalent consumption during the first 24 hours
Time to first analgesic request | Up to 48 hours following surgery
Pain Assessment (VAS) | at 0, 6, 12, 18 and 24 hours
  Visual Analogue Scale(VAS) - Pain:Overall pain assessed at rest and on movement A continuous scale comprised of a 100mm (10cm) horizontal line, anchored by 2 verbal descriptions No Pain to Worst Pain
Risk of opioid-related side effects | Up until one month following nerve block
  nausea, vomiting, pruritus, sedation
Block-related complications | Up until one month following nerve block
  vascular puncture, hematoma formation, intravascular injection, epidural anesthesia-bilateral sensory block
Satisfaction with pain management | at 24 hours
  A Patient Diary will be completed to assess overall satisfaction with analgesic technique 10 cm scale with "not satisfied at all" and "very satisfied" at either end

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, Principal Investigator — Women's College Hospital

REFERENCES:
- [Background] Kim DH, Beathe JC, Lin Y, YaDeau JT, Maalouf DB, Goytizolo E, Garnett C, Ranawat AS, Su EP, Mayman DJ, Memtsoudis SG. Addition of Infiltration Between the Popliteal Artery and the Capsule of the Posterior Knee and Adductor Canal Block to Periarticular Injection Enhances Postoperative Pain Control in Total Knee Arthroplasty: A Randomized Controlled Trial. Anesth Analg. 2019 Aug;129(2):526-535. doi: 10.1213/ANE.0000000000003794. PMID 30234517